CLINICAL TRIAL: NCT01599897
Title: A Phase 1, Randomized, Dose-escalation Study to Evaluate the Safety and Immunogenicity of the ID93 + GLA-SE Vaccine at Two Dose Levels of the ID93 Antigen and the GLA-SE Adjuvant in Healthy Adults
Brief Title: Phase 1 ID93 + GLA-SE Vaccine Trial in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Aeras (Other); Paul G. Allen Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IDRI-TBVPX-113
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; TB; Pulmonary; Vaccine
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 2 µg ID93 + 2 µg GLA-SE (Experimental): Low dose and antigen and low dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 10 µg ID93 + 2 µg GLA-SE (Experimental): High dose of antigen and low dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 2 µg ID93 + 5 µg GLA-SE (Experimental): Low dose of antigen and high dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 10 µg ID93 + 5 µg GLA-SE (Experimental): High dose of antigen and high dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 2 µg ID93 alone (Active Comparator): Low dose of antigen alone.
  Interventions: Biological: ID93 alone
- 10 µg ID93 alone (Active Comparator): High dose of antigen alone.
  Interventions: Biological: ID93 alone

INTERVENTIONS:
Biological: ID93 + GLA-SE — ID93 antigen and GLA-SE adjuvant. 3 injections at Days 0, 28, and 56.
  Arms: 10 µg ID93 + 2 µg GLA-SE; 10 µg ID93 + 5 µg GLA-SE; 2 µg ID93 + 2 µg GLA-SE; 2 µg ID93 + 5 µg GLA-SE
Biological: ID93 alone — ID93 antigen alone. 3 injections and Days 0, 28, and 56.
  Arms: 10 µg ID93 alone; 2 µg ID93 alone

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and immunogenicity in healthy adult subjects of an investigational vaccine being developed for the prevention of pulmonary tuberculosis. The vaccine, identified as ID93 + GLA-SE, consists of the recombinant four-antigen Mycobacterium tuberculosis recombinant protein ID93 together with the adjuvant GLA-SE.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the written informed consent process prior to start of screening evaluations
* Male or female who is 18 to 45 years of age at the time of randomization
* Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
* Agrees to avoid elective surgery for the full duration of the study
* For female subjects: agrees to avoid pregnancy through Study Day 238. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), condoms or the combination of diaphragm with spermicide
* Has body mass index (BMI) between 19 and 33 (weight/height2) by nomogram at the time of randomization

Exclusion Criteria:

* Acute illness at the time of randomization
* Oral temperature greater than 37.5C (99.5F) at the time of randomization
* Values for any of the following screening laboratory parameters, from blood collected within 15 days prior to randomization, outside the normal ranges per local laboratory parameters: hemoglobin, hematocrit, absolute neutrophil count, absolute lymphocyte count, white blood cell count, electrolytes, ALT, AST, total bilirubin, alkaline phosphatase (ALP), creatinine, BUN, and lipid profile
* Evidence of systemic or local disease process on screening urinalysis
* Evidence of significant active infection
* Positive laboratory test (e.g., QuantiFERON(R)-TB) evidence of Mtb infection at screening
* History of treatment for active or latent tuberculosis infection
* History or evidence of active tuberculosis
* Has received vaccination or immunotherapy with a BCG product at any time prior to randomization
* Shared a residence within the last year prior to randomization with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
* History of or evidence of current hypertension
* History of autoimmune disease or immunosuppression
* Used immunosuppressive medication within 42 days before randomization (inhaled and topical corticosteroids are permitted)
* Received immunoglobulin or blood products within 42 days before randomization
* Received any investigational drug therapy or investigational vaccine within 182 days before randomization, or planned participation in any other investigational study during the study period
* Received investigational Mtb vaccine at any time prior to randomization
* Unable to discontinue current chronic prescription drug therapy including hormone replacement such as thyroxin, insulin, and medications that can be hepatotoxic or toxic to the bone marrow (such as statins) etc (estrogen and progesterone replacement and contraceptives, topical medications, and nasal steroids are acceptable)
* History or laboratory evidence of immunodeficiency state including but not limited to laboratory indication of HIV 1 infection at screening
* History of allergic disease or reactions (such as an allergic reaction to eggs), including eczema, likely to be exacerbated by any component of the study vaccine
* History of allergic reaction to kanamycin-related antibiotics
* Previous medical history that may compromise the safety of the subject in the study, including but not limited to: severe impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy or infantile spasms
* History of positive tuberculin skin test
* Evidence of chronic hepatitis (e.g., hepatitis B core antibody or hepatitis C antibody) at screening
* History of alcohol or drug abuse within the past 2 years or consumes more than 1 (women) or 2 (men) alcoholic beverage(s) per day
* Tobacco or cannabis smoking 3 or more days per week
* History of keloid formation
* Positive urine test for illicit drugs (opiates, cocaine, amphetamines) at screening
* History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine, including axillary lymphadenopathy
* All female subjects: currently pregnant or lactating/nursing; or positive urine pregnancy test during screening or positive urine pregnancy test on the day of study injection
* Received a tuberculin skin test within 3 months (90 days) prior to the time of randomization
* Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing adverse events. | 420 days
  To evaluate the safety and tolerability of 2 or 10 μg of ID93 together with 2 or 5 μg of GLA-SE compared to 2 or 10 µg of ID93 alone following intramuscular administration on Days 0, 28, and 56. The safety assessments will be based on local and systemic reactions, including reported adverse events, changes in laboratory values, and changes in vital signs. The severity and relationship to treatment will be recorded for all adverse events.

SECONDARY OUTCOMES:
Immunogenicity | Days 0, 1, 3, 7, 14, 28, 42, 56, 70, 84, 238
  To assess the immunogenicity of ID93 + GLA-SE compared to ID93 alone by evaluating IgG antibody and T-cell responses to ID93 at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI); Anna Marie Beckmann, PhD, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States

REFERENCES:
- [Derived] Coler RN, Day TA, Ellis R, Piazza FM, Beckmann AM, Vergara J, Rolf T, Lu L, Alter G, Hokey D, Jayashankar L, Walker R, Snowden MA, Evans T, Ginsberg A, Reed SG; TBVPX-113 Study Team. The TLR-4 agonist adjuvant, GLA-SE, improves magnitude and quality of immune responses elicited by the ID93 tuberculosis vaccine: first-in-human trial. NPJ Vaccines. 2018 Sep 4;3:34. doi: 10.1038/s41541-018-0057-5. eCollection 2018. PMID 30210819